CLINICAL TRIAL: NCT03651752
Title: An Open-Label Study to Evaluate DPCP Ointment for the Treatment of Alopecia Areata
Brief Title: DPCP for the Treatment of Alopecia Areata
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was paused/enrollment on hold after 4 screen failed subjects. No further subjects were enrolled, therefore, no data was available to collect/analyze.
Sponsor: University of Minnesota (Other)
Collaborators: National Alopecia Areata Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DERM-2016-25380
Record Dates: First submitted 2018-08-03; First posted 2018-08-29 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — diphenylcyclopropenone; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diphenylcyclopropenone (DPCP) Ointment (Other): All subjects will be administered a sensitization dose of 0.05 mL 0.4% DPCP ointment formulation topically in the inner aspect of the upper right arm at Day -16, and 0.05 mL of four concentrations (0.1, .05, 0.01, 0.005%), prepared through dilutions in the ointment vehicle, topically on the inner aspect of the left thigh at Day -2. The weakest strength that may cause a minimal reaction (DTH skin reaction score of 1+) after two days will be chosen, and 0.75-1 g of that concentration will be applied to the scalp starting at Week 1 and administered subsequently twice a week for 18 weeks
  Interventions: Drug: Diphenylcyclopropenone (DPCP) Ointment

INTERVENTIONS:
Drug: Diphenylcyclopropenone (DPCP) Ointment — All subjects will be administered a sensitization dose of 0.05 mL 0.4% DPCP ointment formulation topically in the inner aspect of the upper right arm at Day -16, and 0.05 mL of four concentrations (0.1, .05, 0.01, 0.005%), prepared through dilutions in the ointment vehicle, topically on the inner aspect of the left thigh at Day -2. The weakest strength that may cause a minimal reaction (DTH skin reaction score of 1+) after two days will be chosen, and 0.75-1 g of that concentration will be applied to the scalp starting at Week 1 and administered subsequently twice a week for 18 weeks

SUMMARY:
This is an open labeled study to determine the response and characteristics, safety and efficacy, of the proprietary DPCP ointment composition as a topical immunotherapeutic agent for the treatment of extensive alopecia areata.

DETAILED DESCRIPTION:
This is an open labeled study to determine the response and characteristics, safety and efficacy, of the proprietary DPCP ointment composition as a topical immunotherapeutic agent for the treatment of extensive alopecia areata.

Up to 10 subjects with 76% to 99% scalp hair loss that, in the opinion of the PI, are eligible for treatment with DPCP will be enrolled. Patients will be recruited from the new and current patient population seen for alopecia areata through the University of Minnesota Medical Center Dermatology Clinic as well as through partnership with the National Alopecia Areata Foundation Clinical Trials Network, and various media outlets.

The products to be evaluated are as follows:

* 0.05 mL of 0.4% DPCP (sensitization dose) applied topically to the inner aspect of the upper right arm. ("Sensitization and Baseline Sample Collection Visit")
* 0.05 mL four dose concentration matrix of DPCP ointment (0.1, 0.05, 0.01, 0.005%) prepared through dilutions in a non-volatile vehicle (applied to the inner aspect of the left upper thigh). ("Dose Determination Visit"; 10-14 days after the Sensitization Visit)If sensitization is not attained after 10 to 14 days, the procedure will be repeated once.

The subject will return 2 days after the Dose Determination Visit, so the PI or co-PI can assess the dose concentration matrix. The weakest strength concentration that caused a minimal reaction will be used throughout the study. 0.75-1 g of the treatment drug will be aThe treatment drug will be applied by the PI, a trained study coordinator, or a staff member of the Clinical Research Unit at the University of Minnesota. Eligible subjects may begin receiving the study drug immediately after enrollment and screening.

The estimated duration of the study is 22 weeks. See Appendix A for the schedule of visits. There will be a total of 42 visits, beginning with a screening visit followed by a single sensitizing dose of study drug at baseline (Day -16) and a dose determination application at Day -2.

Subjects will undergo twice weekly (+/- 2 days) topical applications of an ointment formulation of DPCP during Weeks 1-18. Application will be done twice per week. The drug application will be performed by a board certified dermatologist for the first two treatment visits (Days 0 and 3; Visits 4 and 5), after which a trained member of the Clinical Research Unit staff will apply the drug twice each week (Weeks 2-18; Visits 6-39). The investigator will attend one treatment visit in the Clinical Research Unit each month to evaluate the extent of hair loss and hair growth (Weeks 4, 8, 12, and 16).

Scalp biopsy specimen collection will be performed at baseline (Day -16, Visit 2), three days after the first treatment (i.e., challenge) application (Day 2, Visit 5), three days after the final application (Week 18 +3d, Visit 39) or during treatment when the study subject is determined to have achieved >=50% hair regrowth.

Three scalp biopsy samples will be collected by a board certified dermatologist. When possible, each sample will be taken from a balding area near an area with hair preferably in a non-androgen dependent site of the scalp. One of the three samples will be frozen in OCT for histologic examination and immunohistochemical studies. A second biopsy sample from an adjacent area will be placed in 10% buffered formalin for histologic examination and assessment of inflammation and hair follicle differentiation. The third sample from each area will immediately be placed in RNAlater (Qiagen, Valencia, CA) for cytokine expression analyses.

Peripheral blood collection for the study will include whole blood for serum and obtaining peripheral blood mononuclear cells (PBMCs). All blood samples will be transported to the Dermatology laboratory at the University of Minnesota for immediate processing and storage for additional biomarker studies.

Research coordinators will be involved in patient recruitment, contact, and scheduling. The PI and research coordinators will all be involved in the collection, analysis, and reporting of collected data.

applied in a thin film that covers the entire scalp.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has clinical diagnosis of extensive alopecia areata (76%-99% involvement as determined by SALT score, Appendix B, Part I).
2. Written informed consent and HIPAA authorization have been obtained.
3. Subject is > 18 to years of age.
4. Female subjects of childbearing potential have a negative pregnancy test and agree to use an acceptable, highly effective method of birth control (i.e., failure rate of less than 1% per year) to prevent pregnancy.
5. Subject agrees to comply with protocol requirements and attend all required study visits and is considered to be a good study subject.
6. Subject meets concomitant medication washout requirements

   -

Exclusion Criteria:

1. Subject has <76 or greater than 99% hair loss.
2. Subject is pregnant or lactating.
3. Subject has current controlled or uncontrolled bacterial, viral (with the exception of herpes simplex), fungal, atypical, or opportunistic infection(s).
4. Subject has a history of substance abuse within the past five years.
5. Immunosuppression (history of transplantation, chemotherapy, splenectomy, HIV).
6. Administration of systemic treatment (e.g., Imuran, biologics) that have an immunomodulatory mechanism of action in the preceding 3 months.
7. Previous treatment with DPCP.
8. Application of topical immunomodulating agent in the preceding 6 weeks.
9. Application of topical or intralesional corticosteroids within the past 6 weeks.
10. Systemic (oral, inhaled, or intravenous) administration of corticosteroid or other systemic treatment (i.e., prednisone) with an immunosuppressive mechanism of action within the past 3 months.
11. Use of light treatments (e.g., PUVA, narrow band UVB) in the preceding 6 weeks.
12. Use of Anthralin in preceding 6 weeks.
13. Use of minoxidil, topical or oral, in the preceding 4 weeks.
14. Subject is currently or has undergone systemic therapy for malignancy within the past five years except for adequately treated Squamous Cell Carcinoma (SCC) or Basal Cell Carcinoma (BCC) of the skin.
15. Clinical evidence of secondary skin infection (i.e., folliculitis).
16. Participation in other therapeutic investigational clinical trials within 4 weeks of enrollment.
17. Evidence of anemia, thyroid disease, sarcoidosis or other medical condition that could be adversely affected by participating in the study.
18. Subject has any medical condition that, in the judgment of the Investigator, would jeopardize the subject's safety following exposure to the administered medications.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of MN Department of Dermatology
Locations (1):
- University of Minnesota Department of Dermatology, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diphenylcyclopropenone (DPCP) Ointment
Started | 4
Completed | 0
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Screen failure | 3

BASELINE CHARACTERISTICS:
Arm/Group | Diphenylcyclopropenone (DPCP) Ointment
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Alopecia Areata That Have Increased Hair Growth as Assessed by SALT Score
Description: Efficacy will be assessed as follows; a. Severity of Alopecia tool (SALT) score: Percentage of hair loss on the scalp will be determined using he SALT score, a global alopecia areata severity score based on scalp hair loss. The SALT score is calculated by visually examining four descrete areas of the scalp, measuring the percentage of terminal hair loss in each area. b. Scalp Photograhpy. c. Hair pull tests (positive or negative)
Time Frame: 18 weeks
Population: The study was paused/enrollment on hold after 4 screen failed subjects, including 1 AE. No further subjects were enrolled, therefore, no data was available to collect/analyze for each outcome.
Arm/Group | Diphenylcyclopropenone (DPCP) Ointment
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Safety will be monitored for side effects at each visit. Adverse events will be tracked for each subject from the time of the first sensitization dose application of the drug until the subject completes the study. Adverse events will be assessed for severity by the investigator and graded on a four point scale: mild, moderate, severe, or life-threatening
Time Frame: 18 weeks
Population: as for outcome 1
Arm/Group | Diphenylcyclopropenone (DPCP) Ointment
Number analyzed (Participants) | 0

3. Secondary Outcome: Determine the Best Starting Dose Range for Future Studies
Description: Dose determination will be assessed utilizing the Immuno Therapeutic Response Skin Reaction Scale (0-4+) with each dose dilution (.1%-.005%) placed every 72 hours on a different skin region. Biopsies will be obtained to identify scalp skin biomarker profiles that characterize a response to DPCP treatment, enabling future potential for predicting individual responses to treatment and the likelihood of a sustained response.
Time Frame: 18 weeks
Population: as for outcome 1
Arm/Group | Diphenylcyclopropenone (DPCP) Ointment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Diphenylcyclopropenone (DPCP) Ointment
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diphenylcyclopropenone (DPCP) Ointment (N=4)
Inflammatory Reaction (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT03651752/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT03651752/ICF_001.pdf